CLINICAL TRIAL: NCT02532387
Title: Outpatient Treatment of Pulmonary Embolism and Deep Vein Thrombosis: Impact of a New Protocol on Emergency Department Efficiency and Patient Safety
Brief Title: Outpatient Treatment of PE and DVT in the Emergency Department
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Christopher Kabrhel, Attending Physician, Massachusetts General Hospital
Other Study IDs: 2015P000877
Record Dates: First submitted 2015-08-20; First posted 2015-08-25 (Estimated); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Pulmonary Embolism; Deep Vein Thrombosis
MeSH Terms: conditions — Pulmonary Embolism; Venous Thrombosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- MGH ED/EDOU patients: Subjects who present to the Massachusetts General Hospital (MGH) ED or EDOU who meet all inclusion and no exclusion criteria.
  Intervention: Telephone follow-up at 7 and 30 days.
  Interventions: Other: Telephone follow-up
- BWH ED/EDOU patients: Subjects who present to the Brigham and Women's Hospital (BWH) ED or EDOU who meet all inclusion and no exclusion criteria.
  Intervention: Telephone follow-up at 7 and 30 days.
  Interventions: Other: Telephone follow-up
- Control subjects: 1. Contemporary controls: subjects diagnosed with Venous Thromboembolism (VTE) in the ED and who are not eligible for outpatient treatment
  2. Historical controls:
     1. Subjects enrolled in the prospective and retrospective SPEED-D study (PI: Kabrhel) and diagnosed with PE between 2006-2012.
     2. Subjects diagnosed with VTE in the MGH and BWH ED in the 18 months prior to the use of the clinical outpatient treatment of PE protocol.

INTERVENTIONS:
Other: Telephone follow-up — Prospectively enrolled subjects will have a 7- and 30-day phone call.
  Groups: BWH ED/EDOU patients; MGH ED/EDOU patients

SUMMARY:
Standardize the approach to outpatient Pulmonary Embolism (PE) and Deep Vein Thrombosis (DVT) treatment.

DETAILED DESCRIPTION:
In the current protocol, we will study the outcomes most likely to influence emergency physician behavior, such as improved Emergency Department (ED) throughput, and decreased ED and Emergency Department Observation Unit (EDOU) length of stay. Metrics such as decreased admissions are also very important to hospital administrators so our results will have impact outside the ED as well. At the end of this study we will demonstrate that a carefully planned and data-driven approach to the outpatient treatment of Pulmonary Embolism (PE) is safe, improves operational metrics, and reduces cost.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 years of age or older at time of enrollment.
* Subject is diagnosed with acute VTE (DVT or PE) in the MGH or BWH ED or transferred to the MGH or BWH ED (e.g from a clinic or outside hospital) with a diagnosis of acute VTE.
* Subject is treated as an outpatient (i.e. discharged) directly from the ED or admitted to the ED Observation Unit/ED Short Stay Unit on the outpatient treatment protocol.

Exclusion Criteria:

* Subjects admitted from the ED to an inpatient service will not be enrolled as study subjects, but will be used as contemporary controls.
* Subjects who are unable to understand or provide informed consent.
* Subjects unable or unlikely to follow up (e.g. prisoners).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a multi-center prospective, observational study of MGH or BWH patients with PE or DVTwith historical and contemporary controls.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Efficiency & cost of clinical protocol | Up to 30 days
  To compare patients diagnosed with VTE after protocol implementation to those diagnosed with VTE prior to protocol implementation in terms of four measures of efficiency:
  A) ED length of stay - defined as time from ED registration to departure from the ED (to either the inpatient floor or to the EDOU).
  B) ED disposition time - defined as time from ED registration to bed request.
  C) Hospital length of stay - defined as time from ED registration to departure from the hospital.
  D) Cost - defined as the estimated cost of care including diagnostic testing, imaging, hospital inpatient/observation unit stay, medication/pharmacy costs.
Safety of clinical protocol | Up to 30 days
  To assess the safety of outpatient VTE treatment, specifically with regards to:
  A) recurrent venous thromboembolism;
  B) bleeding (major or minor);
  C) unscheduled return to hospital for any reason;
  D) death from any cause: occurring up to 30 days after their discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Kabrhel, MD MPH, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts